CLINICAL TRIAL: NCT04008706
Title: A Phase 3b, Multicenter, Open-Label, Single-Arm Study of Acalabrutinib (ACP-196) in Subjects With Chronic Lymphocytic Leukemia.
Brief Title: Acalabrutinib Safety Study in Untreated and Relapsed or Refractory Chronic Lymphocytic Leukemia Patients
Acronym: ASSURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00008; 2019-001573-89 (EudraCT Number)
Record Dates: First submitted 2019-06-19; First posted 2019-07-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; Acalabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: This is a single arm study in which participants will be enrolled into 3 cohorts. In the treatment-naive (TN) cohort, a minimum of 300 participants with treatment-naïve chronic lymphocytic leukemia will be enrolled. In the relapsed/refractory (R/R) cohort, approximately 200 participants with relapsed/refractory chronic lymphocytic leukemia will be enrolled. In the prior ibrutinib cohort, up to 40 participants with Prior ibrutinib therapy will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib (Experimental): Participants will be enrolled into 3 cohorts. In the treatment-naive cohort, a minimum of 300 participants with treatment-naïve chronic lymphocytic leukemia will be enrolled. In the relapsed/refractory cohort, approximately 200 participants with relapsed/refractory chronic lymphocytic leukemia will be enrolled. In the prior ibrutinib cohort, approximately 40 participants with Prior ibrutinib therapy will be enrolled.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib will be administered as one 100 mg capsule taken orally, twice daily with 8 ounces (approximately 240 mL) of water.
  Other Names: ACP-196

SUMMARY:
This is a global, Phase IIIb, multicenter, open-label, single-arm study to evaluate the safety and efficacy of acalabrutinib 100 mg twice daily (bid) in approximately 540 participants with chronic lymphocytic leukemia (CLL). Participants will be enrolled into 3 following cohorts: treatment-naive (TN), relapsed/refractory (R/R), and prior ibrutinib therapy. For this study, participants in the UK will be enrolled ONLY into the R/R cohort or the prior ibrutinib cohort. Participants in the US will be enrolled ONLY into the TN or R/R cohort. Participants will remain on study intervention until completion of 48 cycles (28 days per cycle), or until study intervention discontinuation due to, for example disease progression, or toxicity, withdrawal of consent, loss to follow-up, death, or study termination by the sponsor whichever occurs first. The duration of the study will be approximately 72 months from the first participant enrolled. This duration includes an estimated 24-month recruitment time and an assumed 48 cycles of study intervention (28 days per cycle); additional study time will be accrued during the Disease Follow up period for those participants remaining on study intervention after completion of 48 cycles prior to the final data cutoff (DCO) (the amount of time will vary by participant).

DETAILED DESCRIPTION:
This is a Global, Phase IIIb, multicenter, open-label, single-arm study to evaluate the safety and efficacy of acalabrutinib 100 mg bid in approximately 540 participants with CLL. Participants will be enrolled into one of the 3 following cohorts:

* Treatment-naive (TN): participants who have had no prior treatment for CLL and who have either a score > 6 on the cumulative illness rating scale and/or have a creatinine clearance of 30 to 69 mL/min using the Cockcroft-Gault equation (minimum of 300 participants). This cohort will not be enrolled in the UK.
* Relapsed/refractory (R/R): participants who have received prior treatment for CLL and who have either relapsed or refractory CLL (approximately 200 participants).
* Prior ibrutinib therapy cohort: participants who have received prior ibrutinib for CLL and who discontinued the medication for any reason prior to disease progression (up to 40 participants). This cohort will not be enrolled in the US.

Overall response and progression assessments will be conducted by the investigator in accordance with the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria. Overall response assessments will be based on physical examinations, recording of symptoms, radiologic evaluations, and hematologic evaluations.

Treatment period consists of 48 cycles [each cycle is 28 days). Study medication (acalabrutinib 100 mg bid) will be administered until disease progression, toxicity requiring discontinuation, completion of 48 cycles of study medication, withdrawal of consent, loss to follow-up, death, or study termination by the sponsor, whichever comes first.

48 Cycles: From Cycle 1 to Cycle 6, in-clinic visits will occur every cycle and during each visit, in-clinic assessments will be carried out. From Cycle 7 to Cycle 12, in-clinic visits will occur every 3 cycles and during each visit, in-clinic assessments will be carried out. From Cycle 13 to Cycle 48, in-clinic visits will occur every 3 cycles and in-clinic assessments will be carried out every 6 cycles.

Safety follow up visits will occur approximately 30 days from the last dose of study treatment.

If a participant continues to derive benefit from treatment at the end of 48 cycles prior to the final DCO, they will continue to be provided with study intervention and will be followed in the Disease Follow-up period every 24 weeks (q24w) until study intervention discontinuation due to, for example, disease progression or toxicity, withdrawal of consent, loss to follow-up, death, or study termination by the sponsor, whichever occurs first. Alternatively, at the end of 48 cycles, a participant can decide to switch to commercial off-study acalabrutinib, if available and permitted by local regulations. Post final DCO, 2 options will be considered: participants may be transitioned to another study or may shift to a commercial supply of acalabrutinib/off-study acalabrutinib as permitted by local regulations. Participants who switch to off-study acalabrutinib will be considered as having completed the study and therefore will not have any additional study assessments, including the safety follow-up visit and disease Follow-up period.

The duration of the study will be approximately 72 months from the first participant enrolled. This duration includes an estimated 24-month recruitment time and an assumed 48 cycles of study intervention (28 days per cycle); additional study time will be accrued during the Follow-up period for those participants remaining on study intervention after completion of 48 cycles prior to the final DCO (the amount of time will vary by participant).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place)
2. Diagnosis of CLL that meets all published diagnostic criteria (Hallek et al. 2018):

   1. Monoclonal B-cells (either kappa or lambda light chain restricted) that are clonally co-expressing ≥1 B-cell marker (CD19, CD20, and CD23) and CD5 during screening
   2. Prolymphocytes may comprise <55% of blood lymphocytes during screening
   3. Presence of ≥5 × 10^9 B lymphocytes/L (5000/μL) in the peripheral blood (at any point since the initial diagnosis)
3. Active disease per at least 1 of the following iwCLL 2018 criteria

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin <10 g/dL) and/or thrombocytopenia (platelets <100,000/μL).
   2. Massive (i.e., ≥6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (i.e., ≥10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy
   4. Progressive lymphocytosis with an increase of >50% over a 2-month period or a lymphocyte doubling time (LDT) of <6 months. LDT may be obtained by linear regression extrapolation of absolute lymphocyte count obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In participants with initial blood lymphocyte counts of <30x10^9/L (30,000/μL), LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g., infections) should be excluded.
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy
   6. B-symptoms documented in the participant's chart with supportive objective measures, as appropriate, defined as ≥1 of the following disease-related symptoms or signs: o- Unintentional weight loss ≥10% within the previous 6 months before screening o- Significant fatigue (Eastern Cooperative Oncology Group [ECOG] performance status ≥2; inability to work or perform usual activities) o- Fevers higher than 100.5°F or 38.0°C for ≥2 weeks o- Night sweats for ≥1 month before screening without evidence of infection
4. Must meet one of the following criteria:

   a. Have received no prior therapy for treatment of CLL and meets one of the following criteria (for this study, participants in the UK will be enrolled ONLY in the R/R or the prior ibrutinib cohort): i. A score of >6 on the Cumulative Illness Rating Scale (CIRS) ii. Creatinine clearance of 30 to 69 mL/min using the Cockcroft-Gault equation b. Have previously received therapy for CLL and have either refractory or relapsed CLL c. Have received prior ibrutinib therapy (i.e., defined as a participant who discontinued a ibrutinib for any reason prior to disease progression) for CLL (participants in the US will not be enrolled into the prior ibrutinib therapy cohort)
5. ECOG performance status of ≤2
6. Female participants of childbearing potential (i.e., not surgically sterile or postmenopausal) who are sexually active with a non-sterilized male partner must use ≥1 highly effective method of contraception from the time of screening and must agree to continue using such precautions for 2 days after the last dose of study intervention. Contraception measures and restrictions on sperm donation are not required for male participants.
7. Fluorescence in situ hybridization (FISH) for which the next-generation sequencing (NGS) method is preferred) within 60 days during screening up to before the first dose reflecting the presence or absence of del(17p), del(13q), del(11q), and trisomy of chromosome 12 along with the percentage of cells with the deletion, along with TP53 sequencing. Participants must also have molecular analysis to detect IGHV mutation status (NGS is the preferred method) at screening if not done at any time point before that since diagnosis.
8. Each participant (or legally authorized representative if allowed per local regulations) must be willing and able to adhere to the study visit schedule, understand and comply with other protocol requirements, and provide written informed consent and authorization to use protected health information.

Exclusion Criteria:

1. Participants who have had disease progression while on a BTKi for any malignant or nonmalignant condition
2. Prior malignancy (other than CLL), except for adequately treated basal cell or squamous cell skin cancer, in situ cancer, early stage prostate cancer, or other cancer from which the participant has been disease-free for ≥2 years
3. History of confirmed progressive multifocal leukoencephalopathy
4. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months before screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval using Fridericia's formula (QTcF) >480 msec at screening. Note: Participants with rate-controlled, asymptomatic atrial fibrillation are allowed to enroll in the study (For prior ibrutinib therapy cohort only, except in Finland and the Republic of South Korea, where this is applicable to all 3 cohorts; also, the prior ibrutinib therapy cohort will not be enrolled in the US).
5. Malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
6. Evidence of active Richter's transformation. If Richter's transformation is suspected (i.e., lactate dehydrogenase [LDH] increased, asymmetric fast lymph node growth or clinical suspicion), it should be ruled out with positron emission tomographycomputed tomography (PET-CT) and/or biopsy according to guidelines.
7. Central nervous system (CNS) involvement by CLL.
8. Known history of human immunodeficiency virus, serologic status reflecting active hepatitis B virus or hepatitis C virus infection, any uncontrolled active systemic infection along with participants who are on ongoing anti-infective treatment and participants who have received vaccination with a live attenuated vaccine within 4 weeks before the first dose of study intervention.

   1. Participants who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antibody (anti-HBs) negative will need to have a negative hepatitis B virus PCR result before enrollment. Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B virus PCR positive will be excluded.
   2. Participants who are hepatitis C virus antibody positive will need to have a negative hepatitis C virus PCR result before enroll.lment. Those who are hepatitis C virus PCR positive will be excluded
9. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (>20 mg daily of prednisone or equivalent for longer than 2 weeks).
10. History of stroke or intracranial hemorrhage within 6 months before the first dose of study intervention.
11. History of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
12. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
13. Major surgical procedure within 4 weeks before first dose of study intervention. Note: Participants who have had major surgery must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study intervention.
14. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Participants receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment in this study.
15. All participants requiring or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days before first dose of study intervention. Based on the known metabolic/transport pathways involved in the disposition of acalabrutinib and the commonly known novel oral anticoagulants (eg, apixaban, rivaroxaban, and edoxaban), no clinically relevant interaction is expected following coadministration of these agents.
16. Absolute neutrophil count (ANC) <0.50 x 10^9/L or platelet count <30 x 10^9/L, unless proven due to CLL and raised above the limits by granulocyte colony-stimulating factor (G-CSF) therapy and/or pooled platelet transfusion
17. Total bilirubin >3.0x upper limit of normal (ULN); or aspartate aminotransferase or alanine aminotransferase >3.0x ULN. Exception will be for Gilbert syndrome; if an investigator feels that a participant's total bilirubin is elevated secondary to Gilbert's, the participant must have a documented unconjugated bilirubin being >80% of the total bilirubin number. The investigator must also document that hemolysis has been ruled out along with (near)-normal lactate dehydrogenase and haptoglobin
18. Estimated creatinine clearance of <30 mL/min, calculated using the formula of Cockcroft and Gault or by direct assessment (i.e., creatinine clearance or ethylene diamine tetra-acetic acid (EDTA) clearance measurement)
19. Breastfeeding or pregnant
20. Received any chemotherapy, external beam radiation, investigational drug, or any other anti-CLL therapy within 30 days before first dose of study intervention
21. Concurrent participation in another therapeutic clinical study
22. History of or ongoing interstitial lung disease
23. Requiring long-term (> 1 week) treatment with a strong cytochrome CYP3A inhibitor/inducer. In addition, the use of strong or moderate CYP3A inhibitors or inducers within 7 days of the first dose of study intervention is prohibited.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From screening to safety follow-up period (approximately 30 days from last dose)
  To evaluate the safety and tolerability of acalabrutinib monotherapy in participants with treatment-naïve or relapsed/refractory chronic lymphocytic leukemia.

SECONDARY OUTCOMES:
Overall response (OR) | 1 year after initial dose of study drug
  To evaluate the investigator-assessed OR in participants receiving acalabrutinib monotherapy.
Duration of response (DOR) | The time from the first objective response to the time of documented disease progression or death due to any cause, whichever occurs first within the time period to complete up to 48 cycles of treatment (each cycle is 28 days)
  To evaluate the investigator-assessed DOR in participants receiving acalabrutinib monotherapy.
Progression-free survival (PFS) | The interval from the start of study treatment to completion of 48 cycles (each cycle is 28 days) or the earlier of the first documentation of disease progression or death from any cause
  To evaluate the investigator-assessed PFS in participants receiving acalabrutinib monotherapy.

OTHER OUTCOMES:
Plasma concentrations of acalabrutinib and ACP 5862 | At Day 1 of Cycle 3 and Day 1 of Cycle 15
  To characterize the pharmacokinetics of acalabrutinib and its metabolite (ACP-5862).
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) | Up to 48 cycles (each cycle is 28 days)
  To evaluate participant-reported symptoms and health-related quality of life following treatment with acalabrutinib monotherapy. EORTC QLQ-C30 scale scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 48 cycles (each cycle is 28 days)
  To evaluate participant-reported symptoms following treatment with acalabrutinib monotherapy using PRO-CTCAE. Patient-reported outcomes (PROs), an umbrella term referring to all outcomes and symptoms, are directly reported by the participant. Around 81 symptoms of the CTCAE v4 have been identified to be amenable to participant reporting. These symptoms have been converted to participant terms (e.g., CTCAE term "myalgia" converted to "aching muscles"). For several symptoms, like fatigue and pain, additional questions are asked about symptom frequency (never to almost constantly), severity (none to very severe, and interference with usual activities (not at all to very much). For this study, the following items are considered relevant and will be assessed: headache, diarrhea, fatigue, nausea, vomiting, abdominal pain, rash, muscle pain, nose bleed, heart palpitations, bruising, joint pain, and constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Habib, MD, Study Director — AstraZeneca; Dr. Carsten Niemann, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (93):
- United States (19):
  - Research Site, Chandler, Arizona
  - Research Site, Long Beach, California
  - Research Site, Redlands, California
  - Research Site, Whittier, California
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
- Australia (6):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, Clayton
  - Research Site, Fitzroy
  - Research Site, Nedlands
  - Research Site, South Brisbane
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Odense
  - Research Site, Roskilde
- Finland (3):
  - Research Site, Hus
  - Research Site, Kuopio
  - Research Site, Tampere
- France (6):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Limoges
  - Research Site, Reims
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (5):
  - Research Site, Bayern
  - Research Site, Essen
  - Research Site, Homburg
  - Research Site, Porta Westfalica
  - Research Site, Schwäbisch Hall
- Italy (4):
  - Research Site, Catanzaro
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Siena
- Netherlands (3):
  - Research Site, Arnhem
  - Research Site, Dordrecht
  - Research Site, Utrecht
- Norway (3):
  - Research Site, Bergen
  - Research Site, Oslo
  - Research Site, Trondheim
- Russia (6):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Syktyvkar
- South Korea (3):
  - Research Site, Busan
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Ourense
  - Research Site, Oviedo
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Uppsala
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, Newmarket

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home